CLINICAL TRIAL: NCT06715748
Title: Prospective Study Investigating the Effects of Intense Endurance Exercise on the Heart Muscle and the Effect of Exogenous Ketones on Acute Changes and Recovery of the Heart Muscle.
Brief Title: Effects of Exogenous Ketones on Acute Changes and Recovery of the Heart Muscle After Intense Exercise.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B2432023000008
Record Dates: First submitted 2024-11-18; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Exercise-induced Myocardial Damage; Right Ventricular Diastolic Dysfunction
Keywords: Exercise induced cardiac damage; Exogeneous ketone; Cardiac Recovery; CMR; Cardiac US; Troponine; Lpa; Exercise-CMR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLACEBO (Placebo Comparator): Participants will perform a randomized, double-blind ZWIFT event, once with ketone ester intake and once with placebo, separated by an interval of 1-3 weeks. Ketones and placebo will be orally administered according to a fixed schedule.
  Interventions: Dietary Supplement: Placebo
- Keton (Active Comparator): Participants will perform a randomized, double-blind ZWIFT event, once with ketone ester intake and once with placebo, separated by an interval of 1-3 weeks. Ketones and placebo will be orally administered according to a fixed schedule.
  Interventions: Dietary Supplement: Ketone Monoester (KE)

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KE) — Participants will perform a randomized, double-blind ZWIFT event, once with ketone ester intake and once with placebo, separated by an interval of 1-4 weeks. Ketones and placebo will be orally administered according to a fixed schedule.
  Arms: Keton
Dietary Supplement: Placebo — Participants will perform a randomized, double-blind ZWIFT event, once with ketone ester intake and once with placebo, separated by an interval of 1-3 weeks. Ketones and placebo will be orally administered according to a fixed schedule.
  Arms: PLACEBO

SUMMARY:
It is well known that scar tissue on the heart muscle can cause (life-threatening) arrhythmias. However, the exact cause of this scar tissue is not entirely clear. It is possible that prolonged and intense exercise is associated with (limited) inflammation of the heart muscle, carrying the risk of scar tissue development.

The aim of this project is to evaluate the impact of prolonged and intense exercise on the heart. Participants will be asked to cycle for a total of 3 hours, of which 2 hours will be at an intense pace. Approximately 30 recreational cyclists will be invited to participate in this research project. Specifically, the investigators want to examine whether prolonged and intense exercise is associated with inflammation of the heart muscle and whether it affects heart function recovery. The research project will take place in a laboratory setting, where heart rate, blood pressure, food and fluid intake, and exertion level will be monitored. Before, after and 20-24h after the intense exercise, a lab test and extensive heart imaging will be performed using magnetic resonance imaging (MRI) and cardiac ultrasound. The investigators aim to study the effect of ketone intake (a dietary supplement that may enhance performance or recovery) on recovery. For this, a double blind cross-over design will be setup. Participants will complete the same exercise twice, with a 1-3 week interval, once with a placebo and once with ketones. All the same baseline, post-exercise and recovery investigations will be perfromed.

In the second part of the study, the investigators will evaluate and compare various rhythm-monitoring devices, both during intense exercise and in daily life. For this, participants will be asked to wear each of four devices for one week in a home setting. These are very small devices that are not externally visible when worn under clothing.

Participation in this project will involve a various questionnaires and tests.

DETAILED DESCRIPTION:
### BACKGROUND:

It has already been established that extensive exercise results in functional and biochemical myocardial damage. However, the development of exercise-induced myocardial edema remains unclear. Native T1 and T2 mapping techniques in cardiac magnetic resonance imaging (CMR) are sensitive to detecting pathological myocardial fluid accumulation and thus serve as potential biomarkers for identifying pathological myocardial edema. A pilot study conducted by Ghekiere et al. demonstrated a correlation between elevated troponin release and increased T1 mapping values, as well as right ventricular (RV) dysfunction. The objective of this study is to perform an additional study with 30 participants, using an adapted study protocol to overcome the main limitations of the pilot study and to evaluate the effects of exogeneous ketones on acute cardiac changes and recovery.

---

* OBJECTIVES

This research aims to investigate whether cardiac abnormalities develop following intense exercise and whether these abnormalities recover or persist after 20-24 hours. Specifically, the investigators will examine whether myocardial edema, cardiac dysfunction, or abnormalities in contractile reserve occur after intense exercise. The investigators intend to examine whether the use of ketones influences the occurrence and recovery of these cardiac abnormalities. A pilot study by Ghekiere et al. showed a correlation between exercise-induced troponin release and elevated T1 mapping values, along with RV dysfunction. The goal of this study is to further explore these findings in a larger population. The investigators will evaluate whether extensive exercise is associated with pathological levels of fluid accumulation in the myocardium, potentially indicating pathological myocardial edema. Additionally, the investigators will assess if ventricular dysfunction occurs and whether contractile reserve changes following intense exercise. Finally, the investigators will examine whether previous findings recover or remain 24 hours after intense exercise, as well as any potential differences between men and women, and the influence of intake of ketones. These findings could contribute to research on pathological heart damage and sudden death in professional cyclists and potentially shed light on the effects of ketones on recovery from cardiac injury.

1. The investigators will evaluate whether intense endurance exercise affects the heart muscle.
2. The investigators will evaluate whether any effects persist or disappear after 24 hours.
3. The investigators will evaluate potential differences between placebo and ketone intake.
4. The investigators will evaluate potential differences between male and female participants.

   ### STUDY POPULATION

   The inclusion criteria are healthy recreational male and female cyclists between 18 and 50 years old, who have signed an informed consent form. Female participants who take contraceptives will be included to prevent hormonal fluctuations from affecting the study results. Each participant will undergo a detailed questionnaire on their training history. Participants will be included if they achieve a VO2-max/kg value above P90, corrected for age and sex, based on the reference value by E. Van der Steeg et al.

   Exclusion criteria include cardiovascular, metabolic, or respiratory diseases, participants with cardiovascular risk factors, and any contraindications for maximum exercise or MRI. The investigators expect approximately 30 participants.
   * RECRUITMENT AND INFORMED CONSENT

   Participants will be recruited from the personal networks of the research team as well as through local sports clubs. No pressure will be applied on potential participants. Participation is voluntary, and individuals have the right to decline participation or withdraw at any time without providing a reason, without affecting their relationship with the researcher. Local sports clubs will be contacted via email and social media. Participants will receive study information via email and can ask questions about the study at any time by email or phone. The study will be explained again at baseline, and the informed consent will then be offered for signing. Informed consent will be collected by the research team. Separate forms will be provided for the study-specific procedures, clarifying that the study falls outside standard care, so no billing will occur.

   ---

   ### METHODOLOGY

   This is an interventional prospective crossover study. Participants will be recruited through acquaintances and local sports clubs. All participants will receive information and a questionnaire and must sign an informed consent.

   All participants will undergo an VO2-max test before the intense exercise to calculate aerobic and anaerobic thresholds, including VO2 max. Prior to the intense exercise, a baseline CMR study will be performed at rest with T1 mapping and T2 mapping (SA basal and midventricular and HLA), functional measurements (HLA, VLA, 3CH, and SA for both ventricles), stress measurements (Supine Exercise-CMR), and contrast-enhanced imaging to detect fibrosis. Baseline blood tests (Na, K, Ca, Chl, Mg, Creatinine, RBC + Hct, Hg, WBC, platelets, High sens Troponine I and T, Creatine kinase, Creatine kinase-MB, NT-proBNP, CRP, Estrogen, Testosterone, Lpa, NT-pro ANP, Albumine, Dopamine, GDF-15, serum B hydroxybutyrate, glucose, lactate, and urinalysis) will be taken to assess cardiac biomarkers and hydration status. A baseline Cardiac ultrasound will also be performed with ventricular function calculations and strain analysis.

   Participants will then undergo an extensive exercise session in controlled conditions (temperature and humidity) at a research lab, the Rehabilitation and Health Center (ReGo) of the Jessa Hospital. All participants will complete a standardized route using a ZWIFT setup, a virtual indoor training setup. The route lasts three hours and is individually adjusted based on the anaerobic threshold, aiming to maintain anaerobic exercise for 1.5-2.0 hours. During the test, a bicycle trainer (Wahoo Kickr) will be provided on which participants can mount their own bicycle. Food and fluid intake will be standardized. Heart rate and hydration balance will be monitored before, during and after the exercise. Glucose, lactate and beta-hydroxybutyrate serum levels will be monitored before, during and after the exercise on capillary blood samples.

   Heart rhythm will be continuously monitored before, during, and after exercise using several devices to compare and validate them in both clinical and home settings (devices: Fourth Frontier X2, Byteflies patch, Rooti Rx). All devices have CE marking, are very small and are not externally visible, and have been used in clinical situations. The monitoring setup will avoid disrupting daily activities.

   Participants will perform a randomized, double-blind ZWIFT event, once with ketone ester intake and once with placebo (an isocaloric medium-chain triglyceride composition), separated by an interval of 1-3 weeks. Ketones and placebo will be orally administered according to a fixed schedule.

   Three to six hours post-exercise, all participants will undergo Cardiac ultrasound, CMR examination with the same sequences as the baseline study, blood tests, and urinalysis. The same tests will be repeated 24 hours after baseline. Cardiac ultrasound evaluation will be performed by an experienced cardiologist. CMR post-processing will be conducted by two experienced cardiac radiologists, and rhythm monitoring will be assessed by an experienced cardiologist.

   Medical procedures will be performed by trained nursing staff and physicians according to usual clinical procedures. Rhythm monitoring data will be analyzed anonymously using company-provided software.
   * RISK-BENEFIT BALANCE

     * There is minimal risk associated with intense exercise. In rare cases, intense exertion can trigger arrhythmias. Previous studies have shown that sudden death occurs in about 1-2 cases per 100,000 athletes per year and 1 per 1 to 4 million hours of exercise. The investigators suspect the risk for our participants will be lower, as they will undergo cardiac evaluation before exercise, and the exercise will be conducted in a controlled setting. The controlled environment is likely to reduce the likelihood of serious complications, as potential issues can be identified and treated early.
     * There is a small chance that the tests may reveal abnormalities that would otherwise remain unnoticed and pose no symptoms or danger. Such findings may cause unnecessary worry. If this occurs, the investigators will fully inform participants about the significance. Conversely, potentially early pathological findings with no symptoms may also be identified, allowing for timely assessment and treatment, potentially preventing or improving long-term outcomes.
     * There is a very small risk of an allergic reaction to gadolinium contrast.
   * DATA ANALYSIS

   Basic CMR post-processing will be performed on a commercial workstation used in routine clinical settings. Cine imaging of the heart will be segmented with commercially available software (NeoSOFT, USA). All study data will be pseudonymized.

   Left ventricular (LV) and right ventricular (RV) volumes will be outlined to calculate ejection fraction, end-diastolic volume, end-systolic volume, cardiac index, and cardiac mass. The thickness of the LV lateral wall and septum will be measured on SA and HLA images. Myocardial T1 and T2 relaxation times will be determined. Analyses will be conducted by two independent cardiac radiologists with expertise in cardiac imaging, blinded to all study data.

   Cardiac ultrasound will be performed and analysed by a cardiologists

   Raw ECG data will be made available via software provided by the respective companies (Byteflies, Fourth Frontier, and Rooti) and evaluated by an experience cardiologist.

   Statistical analysis will be conducted using IBM SPSS version 27.0 (IBM SPSS Statistics for Windows, Chicago, IL, USA). A Shapiro-Wilk test will be conducted to test the normal distribution of the data (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* healthy recreational male and female cyclists between 18 and 50 years old, who have signed an informed consent form.
* Participants will be included if they achieve a VO2-max/kg value above P90, corrected for age and sex, based on the reference value by E. Van der Steeg et al.

Exclusion Criteria:

* Cardiovascular, metabolic, or respiratory diseases
* Participants with cardiovascular risk factors
* Contraindications for maximum exercise
* Contraindications for MRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Troponin release after identical strenuous exercise is significant different with Ketone ester supplementation compared to Placebo | All participants will do two identical streneous exercise within two weeks, day 1 with intake of Keton ester and day 2 with intake of Placebo. All participants will recieve baseline, post race and 20-24 hours post baseline investigations.
Change in contractile reserve measured with Exercise-CMR after identical streneous exercise will be significant different with Ketone ester supplementation compared to placebo. | All participants will do two identical streneous exercise within two weeks, day 1 with intake of Keton ester and day 2 with intake of Placebo. All participants will recieve baseline, post race and 20-24 hours post baseline investigations.

SECONDARY OUTCOMES:
20-24h after indentical streneous exercise, recuperation of ventricular contractile reserve measured with Exercise-CMR will be significant different with Ketone ester supplementation compared to placebo. | All participants will do two identical streneous exercise within two weeks, day 1 with intake of Keton ester and day 2 with intake of Placebo. All participants will recieve baseline, post race and 20-24 hours post baseline investigations.
Change in T1-mapping values measured on CMR after identical strenuous exercise is significant different with Ketone ester supplementation compared to Placebo | All participants will do two identical streneous exercise within two weeks, day 1 with intake of Keton ester and day 2 with intake of Placebo. All participants will recieve baseline, post race and 20-24 hours post baseline investigations.
Change in T2-mapping values measured on CMR after identical strenuous exercise is significant different with Ketone ester supplementation compared to Placebo | All participants will do two identical streneous exercise within two weeks, day 1 with intake of Keton ester and day 2 with intake of Placebo. All participants will recieve baseline, post race and 20-24 hours post baseline investigations.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data will be available 3 months after summary data are published
Access Criteria: Data will be available upon request from the principal investigator, who will provide a secure clould solution to acces the data.

REFERENCES:
- [Background] Ghekiere O, Herbots L, Peters B, Berg BV, Dresselaers T, Franssen W, Padovani B, Ducreux D, Ferrari E, Nchimi A, Demanez S, De Bosscher R, Willems R, Heidbuchel H, La Gerche A, Claessen G, Bogaert J, Eijnde BO. Exercise-induced myocardial T1 increase and right ventricular dysfunction in recreational cyclists: a CMR study. Eur J Appl Physiol. 2023 Oct;123(10):2107-2117. doi: 10.1007/s00421-023-05259-4. Epub 2023 Jul 22. PMID 37480391